CLINICAL TRIAL: NCT00957346
Title: Mifepristone and Misoprostol Versus Misoprostol Alone for Mid-trimester Termination of Pregnancy (14-21 Weeks LMP): A Randomized-controlled Double-blinded Trial
Brief Title: Mifepristone and Misoprostol Versus Misoprostol Alone for Mid-trimester Termination of Pregnancy (14-21 Weeks LMP)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.3.2
Record Dates: First submitted 2009-08-05; First posted 2009-08-12 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Abortion, Induced
Keywords: Pregnancy termination; abortion; medical abortion; 2nd trimester; mifepristone; misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mifepristone + Misoprostol (Experimental): 200 mg mifepristone followed by 400 mcg buccal misoprostol repeated every 3 hours until complete abortion or maximum of 5 doses.
  Interventions: Drug: Mifepristone+misoprostol
- Misoprostol (Placebo Comparator): Placebo resembling 200mcg mifepristone followed by 400 mcg buccal misoprostol repeated every 3 hours until complete abortion or maximum of 5 doses
  Interventions: Drug: Placebo+Misoprostol

INTERVENTIONS:
Drug: Mifepristone+misoprostol — single dose of 200 mg mifepristone followed 24 hours later by 400 mcg misoprostol administered buccally and repeated every 3 hours for a maximum of 5 doses.
  Arms: Mifepristone + Misoprostol
Drug: Placebo+Misoprostol — placebo resembling mifepristone followed 24 hours later by 400 mcg buccal misoprostol repeated every 3 hours until complete abortion or maximum of 5 doses.
  Arms: Misoprostol

SUMMARY:
The primary goal of this study is to determine the clinical advantage of pre-treatment with mifepristone in second trimester misoprostol induction abortion. This will be a randomized controlled double-blinded trial of 20 women comparing misoprostol alone to mifepristone plus misoprostol for second trimester (14-21 weeks' LMP) medical abortion.

ELIGIBILITY:
Inclusion Criteria:

* Meet legal criteria to obtain abortion
* Present with closed cervical os and no vaginal bleeding
* Live fetus at time of presentation for service
* Have no contraindications to study procedures, according to provider
* Be able to consent to procedure, either by reading consent document or by having consent document read to her
* Be willing to follow study procedures

Exclusion Criteria:

* Known previous transmural uterine incision
* Known allergy to mifepristone or misoprostol/prostaglandin or other contraindications to the use of mifepristone or misoprostol
* Any contraindications to vaginal delivery, including placenta previa
* Presentation in active labor (defined as moderate to severe contractions every 10 minutes or less)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Rate of successful abortion: defined as complete evacuation of uterus using study drug without recourse to any additional intervention. | every 3 hours
Induction-to-abortion interval: defined as time elapsed between administration of the first misoprostol dose until expulsion of the fetus; approximately 10-24 hours. | 48 hours

SECONDARY OUTCOMES:
Provision of additional interventions to manage excessive blood loss. | Within 30 days of mifepristone administration.
Total dose of misoprostol. | Assessed at time of complete abortion with study drug alone or when total maximum dose given: approximately 10-24 hours after first dose of misoprostol administration.
Any heavy bleeding, uterine rupture, or infection requiring additional treatment | Within 30 days of mifepristone administration.
Pain experienced by the woman | Assessed during exit interview: approximately 48 hours after first dose of misoprostol administration.
Women's acceptability of the assigned method | Assessed during exit interview: approximately 48 hours after first dose of misoprostol administration.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winkoff, M.D., M.P.H, Principal Investigator — Gynuity Health Projects; Yari Vale-Moreno, M.D., Principal Investigator — University of Puerto Rico Department of Obstetrics and Gynecology; Melanie Pena, MPH, MA, Study Director — Gynuity Health Projects
Locations (1):
- University of Puerto Rico, University District Hospital Medical Science Campus, San Juan, Puerto Rico